CLINICAL TRIAL: NCT06776445
Title: Efficacy and Safety of Different Dose Regimens of Gabapentin for Treating Erythema/Flushing in Rosacea: A Randomized Controlled Trial
Acronym: Gabapenti
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Bin Wei, Director, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2024MSXM069; CSTB2023NSCQ-MSX0078 (Other Grant/Funding Number: Natural Science Foundation of Chongqing, China General Project); 2024MSXM069 (Other Grant/Funding Number: Joint project of Chongqing Health Commission and Science and Technology Bureau)
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Rosacea; Rosacea Subtype 1 (Erythematotelangiectatic)
Keywords: rosacea
MeSH Terms: conditions — Rosacea | interventions — Hydroxychloroquine; Gabapentin; BID protein, human

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- minocycline combined with hydroxychloroquine (Experimental)
  Interventions: Drug: minocycline combined with hydroxychloroquine
- gabapentin 300mg bid (Active Comparator)
  Interventions: Drug: gabapentin 300mg bid
- gabapentin 300mg tid (Active Comparator)
  Interventions: Drug: gabapentin 300mg tid

INTERVENTIONS:
Drug: minocycline combined with hydroxychloroquine — Patients with rosacea were collected and randomly divided into three groups for treatment, one group was treated with minocycline combined with hydroxychloroquine, one group was treated with gabapentin 300mg Bid, and the other group was treated with gabapentin 300mg tid. Before treatment, 4 weeks after treatment, and 8 weeks after treatment, the patient's condition score was statistically analyzed, and the efficacy and difference of each group were observed
  Arms: minocycline combined with hydroxychloroquine
Drug: gabapentin 300mg bid — Patients with rosacea were collected and randomly divided into three groups for treatment, one group was treated with minocycline combined with hydroxychloroquine, one group was treated with gabapentin 300mg Bid, and the other group was treated with gabapentin 300mg tid. Before treatment, 4 weeks after treatment, and 8 weeks after treatment, the patient's condition score was statistically analyzed, and the efficacy and difference of each group were observed
  Arms: gabapentin 300mg bid
Drug: gabapentin 300mg tid — Patients with rosacea were collected and randomly divided into three groups for treatment, one group was treated with minocycline combined with hydroxychloroquine, one group was treated with gabapentin 300mg Bid, and the other group was treated with gabapentin 300mg tid. Before treatment, 4 weeks after treatment, and 8 weeks after treatment, the patient's condition score was statistically analyzed, and the efficacy and difference of each group were observed
  Arms: gabapentin 300mg tid

SUMMARY:
The goal of this clinical trial is to learn if Gabapentin works to treat flushing/erythema associated with rosacea. It will also learn about the safety of drug Gabapentin. The main questions it aims to answer are:

* Does drug Gabapentin reduce flushing and erythema associated with rosacea?
* What medical problems do participants have when taking drug Gabapentin? Researchers will compare Gabapentin to a positive control (minocycline plus hydroxychloroquine, a first-line treatment for rosacea) to see if drug Gabapentin works to reduce flushing and erythema associated with rosacea

ELIGIBILITY:
Inclusion Criteria:

* Initial treatment in our hospital; ② Diagnosed by two experienced dermatologists and in accordance with the updated diagnostic criteria of the National Rosacea Society (NRS) Expert Committee [38], unconscious disorder and no communication disorder; ③ did not receive any other form of treatment within 4 weeks; ④ Patients who were followed up for 8 weeks or more and had complete clinical data; ⑤ Informed consent was signed before treatment, and the clinical data were agreed to be used for scientific research

Exclusion Criteria:

① received other treatment within 4 weeks of this treatment; ② facial flushing caused by other diseases and local irritation; ③ Patients with contraindication to minocycline, hydroxychloroquine, gabapentin and carvedilol; ④ Unable to complete follow-up and serum specimen collection; ○5 patients were intolerant to minocycline, hydroxychloroquine and carvedilol; ○6 Lactation, pregnancy, liver and kidney dysfunction, psychiatric diseases, cardiovascular and cerebrovascular diseases, systemic lupus erythematosus and other systemic diseases.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
the score of CEA ( Clinician Erythema Assessment ) | 4 weeks, 8 weeks, 12 weeks after treatment
  The reduction of the CEA score was compared before treatment, 4 weeks and 8 weeks, 12 weeks after treatment. The CEA score was assessed by a scale, 0 = clear, 1= almost clear, 2 =Mild, 3= Moderate,4= Severe.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Chongqing Medical University, Chongqing, China

REFERENCES:
- [Result] Del Rosso JQ, Webster G, Weiss JS, Bhatia ND, Gold LS, Kircik L. Nonantibiotic Properties of Tetracyclines in Rosacea and Their Clinical Implications. J Clin Aesthet Dermatol. 2021 Aug;14(8):14-21. Epub 2021 Aug 1. PMID 34840653
- [Result] Ma G, Zhang Y, Gao Q, Yuan X, Zhou Z, Jian D, Zhao Z, Wang B, Li J. Gabapentin improves the flushing of rosacea, but not other rosacea symptoms or quality of life: Results from a multicenter, randomized, double-blind, placebo-controlled pilot study. J Am Acad Dermatol. 2025 Apr;92(4):920-922. doi: 10.1016/j.jaad.2024.12.003. Epub 2024 Dec 15. No abstract available. PMID 39681269
- [Result] Wei J, Wan M, Chen Q, Fu J, Yang L, Ni R, Ge L, Dan Y, Chen X, Kong M, Li L, Chen S, Yang S, Zhang L, Xia A, Tang L, Zhang Y, Zhang M, Song Z, Li J. Gabapentin is an efficacy treatment for facial flushing and erythema of erythematotelangiectatic rosacea: A randomized clinical noninferiority trial. J Am Acad Dermatol. 2025 Apr;92(4):927-930. doi: 10.1016/j.jaad.2024.12.011. Epub 2024 Dec 20. No abstract available. PMID 39710117
- [Result] Logger JGM, Olydam JI, Driessen RJB. Use of beta-blockers for rosacea-associated facial erythema and flushing: A systematic review and update on proposed mode of action. J Am Acad Dermatol. 2020 Oct;83(4):1088-1097. doi: 10.1016/j.jaad.2020.04.129. Epub 2020 Apr 29. PMID 32360760
- [Result] Husein-ElAhmed H, Steinhoff M. Evaluation of the efficacy of subantimicrobial dose doxycycline in rosacea: a systematic review of clinical trials and meta-analysis. J Dtsch Dermatol Ges. 2021 Jan;19(1):7-17. doi: 10.1111/ddg.14247. Epub 2020 Sep 28. PMID 32989925
- [Result] Clanner-Engelshofen BM, Bernhard D, Dargatz S, Flaig MJ, Gieler U, Kinberger M, Klovekorn W, Kuna AC, Lauchli S, Lehmann P, Nast A, Pleyer U, Schaller M, Schofer H, Steinhoff M, Schwennesen T, Werner RN, Zierhut M, Reinholz M. S2k guideline: Rosacea. J Dtsch Dermatol Ges. 2022 Aug;20(8):1147-1165. doi: 10.1111/ddg.14849. Epub 2022 Aug 5. PMID 35929658
- [Result] Tu KY, Jung CJ, Shih YH, Chang ALS. Therapeutic strategies focusing on immune dysregulation and neuroinflammation in rosacea. Front Immunol. 2024 Jul 29;15:1403798. doi: 10.3389/fimmu.2024.1403798. eCollection 2024. PMID 39136023
- [Result] Barakji YA, Ronnstad ATM, Christensen MO, Zachariae C, Wienholtz NKF, Halling AS, Maul JT, Thomsen SF, Egeberg A, Thyssen JP. Assessment of Frequency of Rosacea Subtypes in Patients With Rosacea: A Systematic Review and Meta-analysis. JAMA Dermatol. 2022 Jun 1;158(6):617-625. doi: 10.1001/jamadermatol.2022.0526. PMID 35385049